CLINICAL TRIAL: NCT01852552
Title: Costs, Cognitive Abilities and Quality of Life After Transcatheter Aortic Valve Implantation and Surgical Aortic Valve Replacement
Acronym: CCQ
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: Ministry of Health, Italy (Other Government); Region Emilia-Romagna, Italy (Unknown)
Responsible Party: Principal Investigator, Francesco Saia, MD, PhD, Dr., IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: GR-2009-1578270
Record Dates: First submitted 2013-05-08; First posted 2013-05-13 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Aortic Valve Stenosis
Keywords: Aortic stenosis; Transcatheter aortic valve implantation; Aortic valve replacement; Costs; Cognitive function; Quality of life
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Transcatheter aortic valve implantation: All consecutive patients undergoing TAVI at participating centres during study period
  Interventions: Device: transcatheter aortic valve implantation
- Aortic Valve Replacement: All consecutive patients aged ≥ 80 years or with Logistic Euroscore≥ 15% undergoing AVR for AS at participating centers during the period of enrollment
  Interventions: Procedure: Aortic Valve Replacement

INTERVENTIONS:
Device: transcatheter aortic valve implantation — Patients undergoing TAVI with transfemoral, transapical, or any other vascular access
  Other Names: Edwards Sapien XT; Corevalve; Acurate-TA
  Groups: Transcatheter aortic valve implantation
Procedure: Aortic Valve Replacement — Surgical AVR, with all kind of commercially available prosthesis (stented, stentless, mechanical)
  Groups: Aortic Valve Replacement

SUMMARY:
Multicenter, prospective, observational study in aortic stenosis (AS) patients undergoing transcatheter aortic valve implantation (TAVI) or high-risk patients undergoing aortic valve replacement (AVR).

The objectives of the study are:

1. Description of neurocognitive status before and after transcatheter aortic valve implantation and aortic valve replacement procedures
2. Description of Quality of Life (QoL) after these procedures
3. Defining the relevance of baseline psychological, emotional and cognitive factors on the outcomes associated to the different treatment modalities
4. Assessment of costs associated to each of the above mentioned strategies of treatment, including costs of the index hospitalization and costs of follow-up.

DETAILED DESCRIPTION:
In Italy, a nation-wide observational study endorsed by the Superior Institute of Health has been previously launched in order to evaluate appropriateness and effectiveness of aortic valve replacement (AVR) and transcatheter aortic valve implantation (TAVI) procedures: the OBservational Study of Effectiveness of AVR-TAVI procedures for severe Aortic steNosis Treatment (OBSERVANT). The present study was designed to complement the national survey on TAVI and AVR procedures including data about costs, cognitive functions and quality of life after these procedures. This integrated framework may help defining the relevance of baseline psychological, emotional and cognitive factors on the outcomes associated to the different treatment modalities and, on the other hand, should enable accurate evaluation of the impact of each kind of treatment on quality of life and neuropsychological functions. These elements could also represent relevant keys to decision-making to the different therapeutic strategies. In addition, we aim to ascertain costs associated to each of the above mentioned strategies of treatment, including costs of the index hospitalization and follow-up costs. Costs estimate, combined to the integrated physical and mental health status outcome for each treatment modality, may represent the background for subsequent cost-effectiveness analyses.

All consecutive patients undergoing transcatheter aortic valve implantation or aortic valve replacement (if age ≥ 80 years or Logistic Euroscore ≥ 15%) for aortic stenosis at participating centers during the period of enrollment will be included in the registry, after release of written informed consent. Allocation of patients to different treatment groups will be performed jointly by a cardiologist and a cardiac surgeon on the basis of a complete clinical framework, independently from the present study and in accordance with available guidelines. Type of treatment (for example, access site for TAVI, type of prosthesis…) will be decided by the physicians based on local clinical practice and general principles of good clinical practice.

The administration of neurocognitive and quality of life questionnaires will be performed before the procedure and after 3 months and 1 year by trained personnel following standard operation procedures defined by a coordinating unit. A telephone and web-based support for operators will be available throughout the entire duration of the study. A common methodology for data collection and analysis is defined to guarantee data reliability and homogeneity of assessments among the participating units. The cost analysis will be coordinated by the Regional Healthcare and Social Agency of the Emilia Romagna Region.

Data will be collected in a web-based database (OBSERVANT) through dedicated Case Records Forms and a final database will be built by merging this database with a separate database for costs and Hospital Discharge Records and Mortality Registry databases.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients undergoing TAVI at participating centers during the period of enrollment
* All consecutive patients aged ≥80 years or with Logistic Euroscore ≥15% undergoing AVR at participating centers during the period of enrollment

Exclusion Criteria:

* Absence of informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients undergoing TAVI or AVR for AS at participating centers during the period of enrollment
Sampling Method: Non-Probability Sample
Enrollment: 518 (Actual)
Dates: Start 2011-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Mini Mental State Examination (MMSE) | baseline, 3-month, 12-month
  Changes in cognitive function after transcatheter aortic valve implantation and surgical aortic valve replacement
Hospital Anxiety and Depression Scale (HADS) | baseline, 3-month, 12-month
  Changes of emotional status after transcatheter aortic valve implantation and surgical aortic valve replacement
Minnesota Living with Heart Failure Questionnaire (MLHFQ) | baseline, 3-month, 12-month
  Changes in quality of life after transcatheter aortic valve implantation and surgical aortic valve replacement
In-hospital costs | Participants will be followed for the duration of hospital stay, an expected average of 10 days for transcatheter aortic valve implantation and 2 weeks for surgical Aortic Valve Replacement
  Calculation of precise hospital costs for transcatheter aortic valve implantation and surgical Aortic Valve Replacement, including costs of hospitalization, drugs and devices.

SECONDARY OUTCOMES:
Myocardial infarction | 30-day, 12-month and up to 2-year (longest available follow-up)
  Incidence of myocardial infarction
Stroke | 30-day, 12-month and up to 2-year (longest available follow-up)
  Incidence of stroke
Pace-maker implantation | 30-day, 12-month
  Need for permanent pacing
Vascular complications | 30-day
  Incidence of vascular complications as defined by the VARC
Bleedings | 30-day
  Incidence of bleedings as defined by the VARC
Acute kidney injury | 30-day
  Incidence of AKI as defined by the VARC
Follow-up costs | 12-month
  Evaluation of costs during follow-up, including new hospital admissions, outpatient clinic and drugs

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Cardiology, Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy